CLINICAL TRIAL: NCT04488835
Title: A Comparative Study Between Pulsed Electromagnetic Field Therapy and Transcutaneous Electrical Nerve Stimulation in Management of Post-herpetic Neuralgia of the Sciatic Nerve
Brief Title: Pulsed Electromagnetic Field Therapy Versus Transcutaneous Electrical Nerve Stimulation in on Post-herpetic Neuralgia of the Sciatic Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Eid, assistant professor of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 68mm
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Neuralgia,Postherpetic
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS Therapy Group (Experimental): patients in this group received TENS therapy in addition to routine physical therapy
  Interventions: Other: Electromagnetic field therapy and transcutaneous electrical nerve stimulation
- PEMFT group (Experimental): patients in this group received PEMFT therapy in addition to routine physical therapy
  Interventions: Other: Electromagnetic field therapy and transcutaneous electrical nerve stimulation

INTERVENTIONS:
Other: Electromagnetic field therapy and transcutaneous electrical nerve stimulation — Both groups received conventional physical therapy treatment protocol. Moreover, group (A) has an additional TENS application and group (B) had PEMFS application. TENS and the PEMFT were applied once daily, three times per week for 20 minutes for each session. Assessment performed pre and post intervention using visual analogue scale (VAS) and estimation of the carbamazepine intake (CMI).

SUMMARY:
Background and purpose: Post-herpetic neuralgia (PHN) is the most frequent chronic complication of herpes zoster, resulting in post- infectious severe neuropathic pain. Due to drug resistance severe pain; patients with PHN suffer from reduced physical activities, social and psychological manifestations as well as decrease in the quality of life. The purpose of this research was to evaluate the efficacy of pulsed electromagnetic field therapy (PEMFT) versus transcutaneous electrical nerve stimulation (TENS) in the treatment of post-herpetic neuralgia of the sciatic nerve.

Methods: In an eight weeks period of treatemnt, 52 patients were randomly and equally assigned into two groups. Both groups received conventional physical therapy treatment protocol. Moreover, group (A) has an additional TENS application and group (B) had PEMFS application. TENS and the PEMFT were applied once daily, three times per week for 20 minutes for each session. Assessment performed pre and post intervention using visual analogue scale (VAS) and estimation of the carbamazepine intake (CMI).

ELIGIBILITY:
Inclusion Criteria:

* Age from 30-40 years
* History of herpes zoster more than 90 days
* Visual analogue scale is greater than or equal 5 out on a scale from 0 to 10
* All patients were on pain medication "Carbamazepine"

Exclusion Criteria:

* uncooperative behavior
* Intellectual disability to complete the self-evaluation questionnaires

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
neuralgia | 8 weeks
  Visual analogue scale for pain ,zero indicates no pain ten indicates maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Eid, Ass.prof., Principal Investigator — Cairo University
Locations (1):
- Marwa Eid, Cairo, Egypt